CLINICAL TRIAL: NCT06040034
Title: Comparison of Bolus Intravenous Lidocaine Administration With Continuous Intravenous Lidocaine Against Post-Extubation Cough Incidence in Post-Thyroidectomy Patients
Brief Title: Bolus vs. Continuous IV Lidocaine Against Post-Extubation Cough in Post-Thyroidectomy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-202309.01
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Comparison
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Lidocaine Intravenous Infusion (Active Comparator): Patients were given a loading dose of 1.5 mg/kgBW intravenous lidocaine for 10 minutes before induction of anesthesia using a syringe pump, followed by continuous intravenous administration of 1.5 mg/kgBW/hour lidocaine until 30 minutes before the end of the surgery (when the skin is being sutured by the surgeon) using a syringe pump. Continuous administration of lidocaine was prepared by the research team as 10 cc of 20 mg/cc lidocaine in a 10 cc syringe and 10 cc of 0.9% NaCl in a 10 cc syringe.
  Interventions: Drug: Lidocaine IV
- Bolus Lidocaine Intravenous (Active Comparator): Patients were given a loading dose of 1.5 mg/kgBW intravenous lidocaine for 10 minutes before induction of anesthesia using a syringe pump, followed by intravenous infusion of saline with the same volume until 30 minutes before the end of the surgery (when the skin is being sutured by the surgeon) using syringe pump.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — Lidocaine given as bolus or continuous infusion.

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of lidocaine bolus intravenous administration to lidocaine continuous intravenous administration in post thyroidectomy patients to observe the effect against post-extubation cough. The main questions it aims to answer are:

* Cough incidence on both groups
* Which method is preferable to reduce post-extubation cough incidence

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 and 2
* Thyroidectomy patients in Hasan Sadikin Bandung Hospital

Exclusion Criteria:

* Subjects' refusal
* Had history of drug allergy, specifically lidaocaine
* Had history of asthma or other lung diseases
* Active smoker
* History of arrhythmia
* Bradycardia subjects (<60 beats per minute)
* Pregnant people
* Perioperative upper respiratory tract infusion
* Routinely consume ACE inhibitor / bronchodilators / steroid
* Renal dysfunction
* Liver dysfunction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Post-Extubation Cough Grade | 24 hours post operative
  Cough graded according to the following criteria:
  Grade 0: no cough; Grade 1: mild, only 1 cough; Grade 2: moderate, >1 cough lasting <5 seconds; Grade 3: coughing heavily and continuously for >5 seconds)

SECONDARY OUTCOMES:
Number of participant experiencing tachycardia | 24 hours perioperative
  Tachycardia is defined as heart rate >100 beats per minute
Number of participant experiencing bradycardia | 24 hours perioperative
  Bradycardia is defined as heart rate <60 beats per minute
Number of participant experiencing hypertension | 24 hours perioperative
  Increase of blood pressure >20% from initial blood pressure
Number of participant experiencing hypotension | 24 hours perioperative
  Decrease of blood pressure <20% from initial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Iwan Fuadi, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Ardi Zulfariansyah, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Ignatia K Hallis, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia